CLINICAL TRIAL: NCT01802567
Title: A Feasibility Trial Using Molecular-Guided Therapy for the Treatment of Patients With Relapsed and Refractory Childhood Cancer
Brief Title: Molecular-Guided Therapy for Relapsed and Refractory Childhood Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giselle Sholler (Other)
Collaborators: Dell, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Giselle Sholler, Beat Childhood Cancer Chair, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMTRC008
Record Dates: First submitted 2013-02-26; First posted 2013-03-01 (Estimated); Results first posted 2024-04-26 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Neuroblastoma; Medulloblastoma; Brain Tumors; Rare Tumors
MeSH Terms: conditions — Neuroblastoma; Medulloblastoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Guided Therapy- Pediatric Gene Analysis Platform (Experimental): A total of 48 neuroblastoma, brain tumor, and rare tumor patients who are refractory or relapsed on conventional therapy will be treated. Guided therapy will allow the use of any therapeutic combination (up to 4 agents) provided it includes medications contained in the study report. All patients will be followed for survival, disease response, progression and safety. All patients will be treated according to the discretion of the treating oncologist and study committee (minimum 3 oncologists and one pharmacist). Extent of disease will be measured and assessed for changes throughout the course of the study and at 6-8 week intervals (every 2 cycles).
  Interventions: Device: Guided Therapy- Pediatric Gene Analysis Platform

INTERVENTIONS:
Device: Guided Therapy- Pediatric Gene Analysis Platform — A total of 48 neuroblastoma, brain tumor, and rare tumor patients who are refractory or relapsed on conventional therapy will be treated. Guided therapy will allow the use of any therapeutic combination (up to 4 agents) provided it includes medications contained in the study report. All patients will be followed for survival, disease response, progression and safety. All patients will be treated according to the discretion of the treating oncologist and study committee (minimum 3 oncologists and one pharmacist). Extent of disease will be measured and assessed for changes throughout the course of the study and at 6-8 week intervals (every 2 cycles).
  Other Names: Molecular Guided Therapy

SUMMARY:
The purpose of this study is to test the feasibility (ability to be done) of experimental technologies to determine a tumor's molecular makeup (gene expression profile) and mutations. This technology called the "Pediatric Gene Analysis Platform" includes a genomic report (gene expression profile) and a DNA Mutation Panel Report that are being used to discover new ways to understand cancers and potentially predict the best treatments for patients with cancer in the future.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically proven neuroblastoma, brain tumor, or rare tumor and confirmation of refractory or recurrent disease with histologic confirmation at diagnosis or at the time of recurrence/progression
* Subjects must be age >12 months at enrollment.
* Subjects must be age ≤ 21 years at initial diagnosis.
* Subjects must have measurable disease as demonstrated by residual abnormal tissue at a primary or metastatic site measuring more than 1 cm in any dimension by standardized imaging (CT or MRI); tumor must be accessible for biopsy. Patients with bone marrow only disease expected to be >75% tumor are eligible to enroll.
* Current disease state must be one for which there is currently no known curative therapy
* Lansky or Karnofsky Score must be more than 50
* Subjects without bone marrow metastases must have an ANC > 750/μl
* Adequate liver function must be demonstrated, defined as:

  1. Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age AND
  2. SGPT (ALT) < 10 x upper limit of normal (ULN) for age
* A negative serum pregnancy test is required for female participants of child bearing potential (≥13 years of age or after onset of menses)
* Both male and female post-pubertal study subjects need to agree to use one of the more effective birth control methods during treatment and for six months after treatment is stopped. These methods include total abstinence (no sex), oral contraceptives ("the pill"), an intrauterine device (IUD), levonorgestrol implants (Norplant), or medroxyprogesterone acetate injections (Depo-provera shots). If one of these cannot be used, contraceptive foam with a condom is recommended.
* Informed Consent: All subjects and/or legal guardians must sign informed written consent. Assent, when appropriate, will be obtained according to institutional guidelines. Voluntary consent for optional biology studies will be included.

Exclusion Criteria:

* Subjects who have received any cytotoxic chemotherapy within the last 7 days prior to enrollment and 14 days prior to study treatment start date.
* Subjects who have received any radiotherapy to the primary sample site within the last 14 days (radiation may be included in treatment decision after biopsy).
* Subjects receiving anti-tumor therapy for their disease or any investigational drug concurrently
* Subjects with serious infection or a life-threatening illness (unrelated to tumor) that is > Grade 2 (NCI CTCAE V4.0), or active, serious infections requiring parenteral antibiotic therapy.
* Subjects with any other medical condition, including malabsorption syndromes, mental illness or substance abuse, deemed by the Investigator to be likely to interfere with the interpretation of the results or which would interfere with a subject's ability to sign or the legal guardian's ability to sign the informed consent, and subject's ability to cooperate and participate in the study

Min Age: 13 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-03-04 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Sholler, MD, Study Chair — Beat Childhood Cancer at Atrium Health
Locations (13):
- United States (13):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Rady Children's Hospital, San Diego, California
  - Connecticut Children's Hospital, Hartford, Connecticut
  - Arnold Palmer Hospital for Children- MD Anderson, Orlando, Florida
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Levine Children's Hospital, Charlotte, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Blood and Cancer Center, Austin, Texas
  - Primary Children's Hospital, Salt Lake City, Utah

REFERENCES:
- See also: Beat Childhood Cancer Consortium website — http://www.beatcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: A total of up to 48 evaluable subjects (up to 52 enrolled) with childhood cancer that are refractory to or have relapsed on conventional therapy will be treated with molecular guided therapy.
  Subjects will be evaluated in 3 strata:
  * Stratum 1: 16 subjects with refractory/relapsed neuroblastoma
  * Stratum 2: 16 subjects with relapsed or refractory brain tumors Stratum 3: 16 subjects with refractory or relapsed rare tumors
Period: Overall Study
Arm/Group | Overall Study
Started | 52
Completed | 34
Not Completed | 18
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1
Not completed — Lack of Efficacy | 7
Not completed — Consented but did not start therapy | 7
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Groups:
- Guided Therapy- Pediatric Gene Analysis Platform: A total of 48 pediatric cancer (neuroblastoma, brain tumor, and rare tumor) patients who are refractory or relapsed on conventional therapy will be treated. Guided therapy will allow the use of any therapeutic combination (up to 4 agents) provided it includes medications contained in the study report. All patients will be followed for survival, disease response, progression and safety. All patients will be treated according to the discretion of the treating oncologist and study committee (minimum 3 oncologists and one pharmacist). Extent of disease will be measured and assessed for changes throughout the course of the study and at 6-8 week intervals (every 2 cycles).
  Guided Therapy- Pediatric Gene Analysis Platform: A total of 48 neuroblastoma, brain tumor, and rare tumor patients who are refractory or relapsed on conventional therapy will be treated. Guided therapy will allow the use of any therapeutic combination (up to 4 agents) provided it includes medications contained in the study report. All patients will be followed for survival, disease response, progression and safety. All patients will be treated according to the discretion of the treating oncologist and study committee (minimum 3 oncologists and one pharmacist). Extent of disease will be measured and assessed for changes throughout the course of the study and at 6-8 week intervals (every 2 cycles).
Arm/Group | Guided Therapy- Pediatric Gene Analysis Platform
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 49
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 9.7 [1 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 5
  White | 40
  More than one race | 3
  Unknown or Not Reported | 3
Tumor Type [Count of Participants; unit: Participants] — Subjects will be evaluated in 3 strata:
  Stratum 1: refractory/relapsed neuroblastoma Stratum 2: refractory/relapsed brain tumors Stratum 3: refractory/relapsed rare tumors
  Participants
    refractory/relapsed neuroblastoma | 22
    relapsed or refractory brain tumors | 8
    refractory or relapsed rare tumors | 22

OUTCOME MEASURES:

1. Primary Outcome: Determine Feasibility Using Days From the Date of Biopsy to Date of Start of Treatment
Description: Days to treatment is one data point that will be used in order to determine feasibility. The definition of feasibility for this study will include: "Enrollment onto study, RNA expression profile completed, DNA Mutation Panel completed, genomic analysis and report generation, tumor board held with treatment decision, treatment review completed and start of treatment by 21 days post biopsy/surgical resection date, and then completion of 1 cycle of therapy."
Time Frame: Date from biopsy to completion of 1 cycle of therapy, generally about 30 days
Measure: Mean (Full Range); unit: Days
Groups:
- Stratum 1: Subjects with refractory/relapsed neuroblastoma
- Stratum 2: Subjects with relapsed or refractory brain tumors
- Stratum 3: Subjects with refractory or relapsed rare tumors
Arm/Group | Stratum 1 | Stratum 2 | Stratum 3
Number analyzed (Participants) | 19 | 7 | 18
Days | 12.2 [7 to 21] | 19.9 [14 to 30] | 14.9 [9 to 29]

2. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety
Description: To determine the safety of allowing a molecular tumor board to determine individualized treatment plans
Time Frame: Adverse Events were collected starting with the date of the first dose of study drug until 30 days after last dose of study drug, ongoing related adverse events were continued to be followed until resolution, on average of 3 years.
Population: All subjects that started at least one dose of therapy. Outcome measure was reported as an overall study result, and was not reported by cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Guided Therapy- Pediatric Gene Analysis Platform
Number analyzed (Participants) | 45
Participants | 43

3. Secondary Outcome: Overall Response Rate (ORR) of Participants by the Presence of Radiologically Assessable Disease by Cross-sectional CT or MRI Imaging and/or by MIBG or PET Scans.
Description: To determine the activity of treatments chosen based on Overall response rate (ORR) using RESIST criteria. The assessment of response will include the initial measurable targets and will be performed after cycle 2, then after every other cycle. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI imaging and/or by MIBG or PET scans: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease, At least a 20% increase in the sum of the disease measurements for measurable lesions, Stable Disease, Neither sufficient decrease to qualify for PR or sufficient increase to qualify for PD from study entry. Overall Response (OR) = CR + PR.
Time Frame: Followed until off therapy, generally 3 years
Population: Analyzed population only includes evaluable subjects, defined as subjects that made it to an evaluation time point (scans at end of cycle 2), or had a documented progression of disease prior to evaluation time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum 1 | Stratum 2 | Stratum 3
Number analyzed (Participants) | 17 | 7 | 17
Participants
  Complete Response | 1 | 2 | 2
  Partial Response | 0 | 0 | 1
  Stable Disease | 4 | 0 | 6
  Progressive Disease | 12 | 5 | 8

ADVERSE EVENTS:
Time Frame: Adverse Events were collected starting with the date of the first dose of study drug until 30 days after last dose of study drug, ongoing related adverse events were continued to be followed until resolution, on average of 3 years.
Description: Adverse events were reported as a whole for all subjects that started at least one dose of study therapy and were not reported by individual cohort. 45 subjects started at least one dose of study therapy on this trial, therefore 45 will be the analysis population for adverse events.
Groups:
- Guided Therapy- Pediatric Gene Analysis Platform: A total of 48 pediatric cancer (neuroblastoma, brain tumor, and rare tumor) patients who are refractory or relapsed on conventional therapy will be treated. Guided therapy will allow the use of any therapeutic combination (up to 4 agents) provided it includes medications contained in the study report. All patients will be followed for survival, disease response, progression and safety. All patients will be treated according to the discretion of the treating oncologist and study committee (minimum 3 oncologists and one pharmacist). Extent of disease will be measured and assessed for changes throughout the course of the study and at 6-8 week intervals (every 2 cycles).
  Adverse events were reported as a whole for all subjects that started study therapy and were not reported by individual cohort.
Arm/Group | Guided Therapy- Pediatric Gene Analysis Platform
All-Cause Mortality (participants affected / at risk) | 2/45
Serious Adverse Events (participants affected / at risk) | 21/45
Other Adverse Events (participants affected / at risk) | 43/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guided Therapy- Pediatric Gene Analysis Platform (N=45)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Deydration (Metabolism and nutrition disorders) | 1 (1)
Epistaxis (Vascular disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 5 (5)
Fever (General disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hypertension (General disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Infection, lung (Infections and infestations) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Oral mucocitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guided Therapy- Pediatric Gene Analysis Platform (N=45)
Neutropenia (Blood and lymphatic system disorders) | 21 (21)
Anemia (Blood and lymphatic system disorders) | 16 (16)
Anorexia (Metabolism and nutrition disorders) | 8 (8)
Aspartate Transferase Increase (Hepatobiliary disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Leukopenia (Blood and lymphatic system disorders) | 19 (19)
Epistaxis (Vascular disorders) | 4 (4)
Fatigue (General disorders) | 4 (4)
Fever (General disorders) | 4 (4)
Hypertension (General disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (7)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Infection (Infections and infestations) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 10 (10)
Pain (General disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 7 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-06-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT01802567/Prot_SAP_000.pdf
  • Informed Consent Form (2013-08-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT01802567/ICF_001.pdf